CLINICAL TRIAL: NCT05379816
Title: A Prospective Study of Persistent Pain Induced by Uniportal Video-assisted Thoracic Surgery: Incidence, Diagnosis, and Intercostal Nerve Treatment
Brief Title: Persistent Pain Induced by Uniportal Video-assisted Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202108162RINA
Record Dates: First submitted 2022-05-15; First posted 2022-05-18 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-10

CONDITIONS: Post-thoracotomy Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Conservative management indicates medication treatment. Interventional treatment indicate injection treatment
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative treatment (No Intervention): analgesics are used for PTPS
- Interventional treatment (Active Comparator): perineural injection
  Interventions: Procedure: 5% DW perineural injection

INTERVENTIONS:
Procedure: 5% DW perineural injection — 5% DW perineural injection to intercostal nerve
  Arms: Interventional treatment

SUMMARY:
The investigators investigate the prevalence of PTPS in patients receiving with uniportal video-assisted thoracic surgery (VATS), and early identify neuropathic pain as well as treated with neural protective strategy to target intercostal nerve.

DETAILED DESCRIPTION:
More than 30% of patients have persistent pain after thoracic surgery. Intercostal neuralgia is characterized by neuropathic pain in the distribution of affected intercostal nerve(s) (along the ribs, chest, or abdomen) that commonly manifests as a sharp, aching, radiating, burning, or stabbing pain and may be associated with paresthesia such as numbness and tingling. The pain may be intermittent or constant and typically presents as a band-like pain that is wrapped around the chest and back or in a thoracic dermatomal pattern. Pain may last for a prolonged period and may continue long after the disease process has subsided.

Hypertonic dextrose injection (prolotherapy) is reported to reduce pain, including non-surgical chronic low back pain (CLBP), and subcutaneous injection of 5% dextrose is said to minimize neurogenic pain hyperalgesia and allodynia. The mechanism in both cases is unclear, though a direct effect of dextrose on neurogenic pain has been proposed. This study assessed the short-term analgesic effects of epidural 5% dextrose injection compared with saline for non-surgical CLBP.

Intercostal nerve damage is a suspected pathogenic mechanism for developing post-thoracotomy pain syndrome (PTPS). Video-assisted thoracic surgery (VATS) is a minimally invasive procedure that potentially reduces PTPS. However, there was no specific outcome study for uniportal VATS.

In this study, the investigators investigate the prevalence of PTPS in patients receiving uniportal video-assisted thoracic surgery (VATS), identify neuropathic pain early, and treat it with a neural protective strategy to target intercostal pain nerve.

ELIGIBILITY:
Inclusion Criteria:

* PTPS after single port VATS

Exclusion Criteria:

* abnormal sensation
* can not complete questionnaire
* others cause of pain

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | 3 months
  difference of Numerical rating scale, before and after

SECONDARY OUTCOMES:
Quantitative sensory test | 3 months
  difference of cold, warm, tactile detection threshold, before and after

CONTACTS AND LOCATIONS:
Overall Officials: Wen-ying Lin, Dr., Principal Investigator — National Taiwan University
Locations (1):
- National taiwan university cancer center, Taipei, Taiwan